CLINICAL TRIAL: NCT03191370
Title: Pragmatic Randomised Controlled Trial Assessing the Use of a Simple Distraction Technique to Reduce Discomfort When Performing Transnasal Fiberoptic Laryngoscopy in the ENT Outpatient Clinic
Brief Title: Distraction Technique to Reduce Discomfort of Transnasal Fiberoptic Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Lincolnshire Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 280217ArshadFaisal
Record Dates: First submitted 2017-06-07; First posted 2017-06-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pain
Keywords: pain during laryngoscopy, Flexible nasal endoscopy
MeSH Terms: conditions — Pain | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Local Anaesthetic, no distraction (Active Comparator): Will receive local (co-phenylcaine) anesthetic spray (Local Anesthetics,Topical) as an active comparator without distraction during the procedure.
  Interventions: Drug: Local Anesthetics,Topical
- Local Anaesthetic, with distraction (Experimental): Will receive local (co-phenylcaine) anesthetic spray (Local Anesthetics,Topical) with distraction during the procedure. The simple distraction technique is the experimental intervention.
  Interventions: Other: Simple distraction technique; Drug: Local Anesthetics,Topical
- No Local Anaesthetic without distraction (No Intervention): Will receive no local (co-phenylcaine) anaesthetic spray without distraction during the procedure.
- No Local Anaesthetic, with distraction (Experimental): Will receive no local (co-phenylcaine) anesthetic spray with distraction during the procedure. The simple distraction technique is the experimental intervention.
  Interventions: Other: Simple distraction technique

INTERVENTIONS:
Other: Simple distraction technique — Asking the patient to count backwards from 30 to1 in even numbers whilst the procedure is being performed.
  Arms: Local Anaesthetic, with distraction; No Local Anaesthetic, with distraction
Drug: Local Anesthetics,Topical — Anesthetic spray
  Other Names: Co-phenylcaine
  Arms: Local Anaesthetic, no distraction; Local Anaesthetic, with distraction

SUMMARY:
To compare the effectiveness of reducing discomfort during flexible nasal endoscopy using simple distraction techniques compared to topical anaesthetic spray and a control group that does not receive topical anaesthetic spray or a distraction technique.

DETAILED DESCRIPTION:
In this randomised controlled study patients will be randomly allocated into one of four groups; the first group will receive topical (co-phenylcaine) anaesthetic spray without distraction, the second group will receive topical (co-phenylcaine) anaesthetic spray with distraction, the thirds group will receive no topical (co-phenylcaine) anaesthetic spray without distraction and the fourth group will receive no topical (co-phenylcaine) anaesthetic spray with distraction. The distraction technique that will be employed is counting backwards from 30 to 1 in even numbers only. All flexible nasal endoscopies will be performed by either of the two most senior clinicians involved in the study. The procedure will be carried out in standard outpatient clinic room setting. Post procedural discomfort assessments will be undertaken using a visual analogue scale (VAS). Power calculations shows that >24 patients would result in an adequately powered study (>80%). Data analysis will be undertaken by SPSS and independent T-tests will be performed to assess for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants aged 18+
* Patient requires flexible fiberoptic transnasal laryngoscopy.
* Patient has no preferences in relation to which arm of the study they would like to be in.

Exclusion Criteria:

* Flexible nasal endoscopy not indicated
* Local anaesthetic required for other reasons - e.g. vasoconstrictor effects
* Patient has a clear preference to which group they are randomised to
* Significant sino-nasal disease
* Patient under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Discomfort during procedure | 5 minutes
  Visual analogue discomfort scale

CONTACTS AND LOCATIONS:
Overall Officials: Faisal A Arshad, MRCS, Principal Investigator — United Lincolnshire NHS trust
Locations (1):
- United Lincolnshire Hospitals Trust, Lincoln, Research Manager, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conlin AE, McLean L. Systematic review and meta-analysis assessing the effectiveness of local anesthetic, vasoconstrictive, and lubricating agents in flexible fibre-optic nasolaryngoscopy. J Otolaryngol Head Neck Surg. 2008 Apr;37(2):240-9. PMID 19128620
- [Background] Cain AJ, Murray DP, McClymont LG. The use of topical nasal anaesthesia before flexible nasendoscopy: a double-blind, randomized controlled trial comparing cophenylcaine with placebo. Clin Otolaryngol Allied Sci. 2002 Dec;27(6):485-8. doi: 10.1046/j.1365-2273.2002.00608.x. PMID 12472516
- [Background] Choudhury N, Amer I, Daniels M, Wareing MJ. Audiovisual distraction reduces pain perception during aural microsuction. Ann R Coll Surg Engl. 2013 Jan;95(1):34-6. doi: 10.1308/003588413X13511609955535. PMID 23317724
- [Background] Pothier DD, Raghava N, Monteiro P, Awad Z. A randomized controlled trial: is water better than a standard lubricant in nasendoscopy? Clin Otolaryngol. 2006 Apr;31(2):134-7. doi: 10.1111/j.1749-4486.2006.01173.x. PMID 16620333